CLINICAL TRIAL: NCT03267706
Title: Introducing the Comprehensive Palliative Care Tool in Family Medicine : A Pilot Randomized Controlled Trial
Brief Title: Introducing the Palliative Care Comprehensive Tool in Family Medicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ainsley Moore, Associate Professor of Family Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PaCCT
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Palliative Care; Primary Care; Satisfaction
Keywords: Primary care; Palliative care
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Pilot prospective randomized controlled trial
Who Masked: Participant
Masking Description: Patients and caregivers are blinded as to whether their clinician received training and access to the newly introduced comprehensive palliative care tool. Clinicians delivering care are not blinded to use of the tool, outcome assessors are not blinded to the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative Care Comprehensive Tool (Active Comparator): Clinicians within the study will be randomly assigned and trained on the use of the Palliative Care Comprehensive Tool
  Interventions: Other: Palliative Care Comprehensive Tool
- Usual Care (No Intervention): Clinicians within the study will be randomly assigned to usual palliative care (without the newly introduced tool)

INTERVENTIONS:
Other: Palliative Care Comprehensive Tool — Clinicians assigned to the newly developed Palliative Care Comprehensive Tool will be trained during a 1 hour period on the application of the tool; Including rationale for tool development, objective of the tool and demonstration of the tool in action
  Other Names: PaCCT
  Arms: Palliative Care Comprehensive Tool

SUMMARY:
The purpose of this study is to pilot the introduction of a newly developed palliative care tool to clinicians in a family health team. The intent of the tool is to improve the quality and comprehensiveness of palliative care, which effects caregiver and patient satisfaction with care received, as well as clinician satisfaction with their delivery of care. Tool effectiveness will be evaluated by measuring satisfaction scores of caregivers, patients and clinicians who receive training and access to the tool compared to caregivers, patients and clinicians providing usual care (without the tool). Uptake of the tool and user feedback will be collected

DETAILED DESCRIPTION:
A newly developed tool to guide clinicians in best palliative care practices was developed based on a combination of published tools and consultation with primary care, end users (clinicians). The tool will be introduced as a pilot to clinicians who will receive training on use of the tool and access to the tool within a family health team in Ontario, Canada. The tool will be applied in a controlled study environment that randomly assigns clinicians to one of two groups. One group will receive training and access to the tool and the other group of clinicians will continue to provide usual care.The tool will be evaluated based on validated satisfaction surveys completed by caregivers, patients and clinicians. Satisfaction scores of those randomly assigned to care enhanced by the tool will be compared to those receiving usual care at the beginning and end of the study. Uptake of the tool will be measured, as well as user experience with the tool (feasibility and acceptability)

ELIGIBILITY:
Inclusion Criteria:

* Inclusive sample of all clinicians employed at Stonechurch Family Health Centre
* Inclusive sample of all patients over 18 years of age, registered as palliative within Stonechurch Family Health Centre and who are English speaking

Exclusion Criteria: Patients younger than 18 years of age, patients who are non-English speaking

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Caregiver satisfaction | 3 months
  FAMCARE-2 survey to measure caregiver satisfaction

SECONDARY OUTCOMES:
Patient satisfaction | 3 months
  FAMCARE-P13
Clinician satisfaction | 3 months
  Physician Satisfaction with Aspects of Chronic Care (modified)
User feedback | 3 months
  Acceptability and feasibility of the Palliative Care Comprehensive Tool will be sought using the Clinical Sensibility Questionnaire
Uptake of tool | 3 month
  Tool implementation will be (rate of tool uptake by clinician)

CONTACTS AND LOCATIONS:
Overall Officials: Ainsley Moore, MD, Principal Investigator — Department of Family Medicine McMaster University
Locations (1):
- Stonechurch Family Health Centre, Department of Family Medicine McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share data. Data will be stored on secured facility servers.